CLINICAL TRIAL: NCT00711113
Title: An Open, Prospective Study to Evaluate Implant Stability, Marginal Bone Adaptation and the Survival Rate of Astra Tech Dental Implant System, Fixture Osseospeed™, in Patients With Tooth Loss in the Posterior Maxilla in an Early Loading Protocol.
Brief Title: Study on OsseoSpeed™ Implants Replacing 2-5 Teeth in the Posterior Upper Jaw, Restored With Provisional Teeth Attached 6-7 Weeks Later
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YA-OSS-0001
Record Dates: First submitted 2008-07-07; First posted 2008-07-08 (Estimated); Results first posted 2014-02-07 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-01

CONDITIONS: Jaw, Edentulous, Partially
Keywords: Jaw, Edentulous, Partially (posterior maxilla)
MeSH Terms: conditions — Jaw, Edentulous, Partially; Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Device: OsseoSpeed™

INTERVENTIONS:
Device: OsseoSpeed™ — OsseoSpeed™, all dimensions

SUMMARY:
The purpose of the study is to evaluate Astra Tech Dental Implant System, Fixture Osseospeed™, in patients with tooth loss in the posterior maxilla in an early loading protocol. Primary objectives are implant stability, marginal bone adaptation and survival rate.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* 18 years of age and over
* Edentulous in the posterior maxilla, Kennedy classes I or II. Last natural tooth, or previously restored implant in function is canine or first bicuspid.
* Deemed by the investigator as likely to present an initially stabile implant situation suitable for early loading

Exclusion Criteria:

* Untreated caries and/or periodontal disease of residual dentition
* History of edentulism in the area of implant placement of less than two months
* Current need for pre-surgical bone or soft tissue augmentation in the planned implant area.
* History of pre-surgical bone or soft tissue augmentation, within12 months, in the planned implant area.
* Sinus floor thickness of less than 5 mm, verified by periapical radiographs.
* Any systemic or local disease or condition that would compromise post-operative healing and/or osseointegration
* Need for systemic corticosteroids or any other medication that would compromise post-operative healing and/or osseointegration
* Present alcohol or drug abuse
* Unable or unwilling to return for follow-up visits for a period of 5 years
* Current use of smoking tobacco
* Pregnancy or lactation at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2003-12; Primary Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James T Mellonig, D.D.S., M.S, Principal Investigator — University of Texas
Locations (3):
- United States (2):
  - University of Iowa, College of Dentistry, Dow's Institute for Dental Research, Iowa City, Iowa
  - UTHSCSA, San Antonio, Texas
- Universitetsklinik Mainz, Klinik fur ZMK, Mainz, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- OsseoSpeed: Fixture Osseospeed Implants with diameter of 3.5, 4.0, 4.5 and 5.0 mm and lengths of 8, 9, 11, 13, 15 and 17 mm.
Period: Overall Study
Arm/Group | OsseoSpeed
Started | 47
Completed | 36
Not Completed | 11
Not completed — Lost to Follow-up | 9
Not completed — Implant lost | 2

BASELINE CHARACTERISTICS:
Population: Per protocol analysis presented, this includes implants loaded 0 to 56 days from implant placement (80 implants in 32 patients).
Arm/Group | OsseoSpeed
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 30
  Germany | 2

OUTCOME MEASURES:

1. Primary Outcome: Implant Survival Rate
Description: An implant that has failed to osseointegrate, lost its osseointegration or fractured was considered a failure effective from the date of removal. The survival rate for individual implants was analyzed at each visit. Cumulative implant survival rate was calculated using Kaplan-Meier life-table estimation and reported as percentage of survived implants.
Time Frame: At 5 year follow-up
Population: Per protocol analysis presented, this includes implants loaded 0 to 56 days from implant placement (80 implants in 32 patients), of these three implants failed during the 5 year follow-up period.
Measure: Number; unit: percentage of implants
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed
Number analyzed (Participants) | 32
Number analyzed (Implants) | 80
percentage of implants | 96.25

2. Primary Outcome: Implant Stability
Description: Implant stability was evaluated using Resonance Frequency Analysis (RFA). The RFA value was automatically translated into an Implant Stability Quotient index (ISQ), which runs from 1 to 100. The ISQ value indicates the level of stability. Low values (<60) indicate low stability, medium values (60-70) indicate medium stability and high values (>70) indicate high stability.
Time Frame: At 1 year follow-up
Population: Per protocol analysis presented, this includes implants loaded 0 to 56 days from implant placement (80 implants in 32 patients). At 1-year follow-up, 32 patients were still in the study and thus evaluable for the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed
Number analyzed (Participants) | 32
Number analyzed (Implants) | 80
units on a scale | 68.3 (6.7)

3. Primary Outcome: Marginal Bone Adaptation
Description: Marginal bone adaptation was expressed as the distance from the implant reference point to the most coronal bone-to-implant contact on the mesial and distal side of the implant. Bone adaptation in millimeters at follow-up visit were compared to values obtained Baseline (loading). Positive value indicates bone gain and negative value bone loss.
Time Frame: At baseline (loading) and at 5 year follow-up
Population: Per protocol analysis presented and this includes implants loaded 0 to 56 days from implant placement (80 implants in 32 patients). At 5-year follow-up, 27 patients were still in the study and thus evaluable for the analysis.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed
Number analyzed (Participants) | 27
Number analyzed (Implants) | 68
Millimeter | 0.3 (0.9)

ADVERSE EVENTS:
Arm/Group | OsseoSpeed
Serious Adverse Events (participants affected / at risk) | 3/47
Other Adverse Events (participants affected / at risk) | 0/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OsseoSpeed (N=47)
Heart attack (Cardiac disorders) | 1 (2)
Subdural hematoma (Vascular disorders) | 1 (1)
Blod clot in lower leg (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less